CLINICAL TRIAL: NCT00748891
Title: Exploratory Open-Label, Non-randomised, Single Centre Methodology Study Comparing DCE-CT and DCE-MRI as Markers of Changes in Vascular Activity Mediated by a Positive Control Agent [Cediranib (Recentin™; AZD2171), a Potent Inhibitor of VEGF-driven Angiogenesis] in Patients With Advanced Solid Tumour
Brief Title: DCE CT/MRI Scanning Study in Patients With Solid Tumours (AstraZeneca and Royal Marsden Hospital Imaging Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Dr Nick Botwood BSc, MBBS, MRCP, MFPM, Medical Science DirectoR, RECENTIN, AstraZeneca Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D1330C00003; EDRACT nbr 2007-006251-39
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Cancer
Keywords: Cancer; tumour; advanced sold tumour; imaging; DCE-CT Scan; DCE-MRI scan; Cediranib; Recentin
MeSH Terms: conditions — Neoplasms | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Open label 30mg Cediranib administered once daily during scanning phase and if tolerated by patient, until disease progression
  Interventions: Drug: Recentin (Cediranib)

INTERVENTIONS:
Drug: Recentin (Cediranib) — 30mg once daily, oral dose
  Other Names: Cediranib

SUMMARY:
This study is being carried out in patients with advanced solid tumours to assess which of two different types of imaging scans best measures activity of an experimental drug called Cediranib. The study compares the imaging tests: Dynamic Contrast Enhanced CT (DCE-CT) and Dynamic Contrast Enhanced MRI (DCE-MRI). It looks at which of these scans is the most accurate and best predicts a response to the treatment. Cediranib is thought to work by stopping blood flow to cancers, and both of these scans assess blood flow. Studying the response of cancers by measuring changes in their blood flow may provide useful information that will guide the way we manage cancers in the future.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic tumour which is refractory to standard therapies
* At least one lesion size ≥3cm on in longest diameter suitable for repeat assessment by DCE-CT and DCE-MRI
* Patients must be able to undergo DCE-CT and DCE-MRI scanning procedures
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Patients with hormone refractory prostate cancer (HRPC)
* Patients with a history of poorly controlled high blood pressure
* Ineligibility for MRI scanning or DCE-CT or DCE-MRI scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Percentage change in DCE-MRI and DCE-CT vascular parameters. Comparison between vascular parameters of each imaging modality and between modalities. | DCE-MRI and DCE-CT scans taken at Baseline, Day 7 and Day 28. Comparison between modalities from scans taken on Days -8 and Day-1.
Baseline measurements for DCE-MRI-iAUC60(mMol/sec),Ktrans(min-1),ve,vp,kep(min-1,Enhancing Fraction% DCE-CT-Permeability Surface Product(ml/min/100g),Perfusion(ml/min/100g),Mean Transit Time(sec),Blood Volume (ml/100g),Positive Enhancement Integral(Hus). | DCE-MRI and DCE-CT scans taken at Day -8, Day -1, Day 7 and Day 28

SECONDARY OUTCOMES:
Objective tumour response (RECIST )Progression free survival | RECIST scans within 4 weeks prior to first dose then 8 weekly up to 24 weeks, then 12 weekly thereafter
Baseline and on treatment time-point measurements for iAUC60 (mMol/sec) and Positive Enhancement Integral (Hus) | DCE-MRI and DCE-CT scans taken at Day -8, Day -1, Day 7 and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, MD, Study Director — AstraZeneca, Alderley Park; Johann De Bono, MD, Principal Investigator — Institute of Cancer Research, Royal Marsden Hospital
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Messiou C, Orton M, Ang JE, Collins DJ, Morgan VA, Mears D, Castellano I, Papadatos-Pastos D, Brunetto A, Tunariu N, Mann H, Tessier J, Young H, Ghiorghiu D, Marley S, Kaye SB, deBono JS, Leach MO, deSouza NM. Advanced solid tumors treated with cediranib: comparison of dynamic contrast-enhanced MR imaging and CT as markers of vascular activity. Radiology. 2012 Nov;265(2):426-36. doi: 10.1148/radiol.12112565. Epub 2012 Aug 13. PMID 22891356